CLINICAL TRIAL: NCT01693380
Title: Effectiveness Assessment of Vaccinating Schoolchildren Against Influenza the in São Paulo, 2009
Brief Title: Effectiveness Assessment of Vaccinating Schoolchildren Against Influenza
Acronym: Xo_Gripe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BUTANTAN
Record Dates: First submitted 2012-09-10; First posted 2012-09-26 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Influenza; Acute Respiratory Infection
Keywords: Influenza; Vaccination; Vaccines; Schoolchildren; Effectiveness; Intervention studies; Adolescents; Laboratory Confirmed Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; serogroup C meningococcal conjugate vaccine; Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccine (Experimental): Schoolchildren from 6 to 8 years received two intra-muscular doses of 0.5 ml of inactivated influenza vaccine, of the Southern Hemisphere, 2009.
  Schoolchildren above 8 years received one intra-muscular dose of 0.5 ml of inactivated influenza vaccine, of the Southern Hemisphere, 2009.
  Interventions: Biological: Influenza vaccine
- Control vaccine (Sham Comparator): Schoolchildren received one intra-muscular dose of 0.5 ml of Meningococcal C conjugate vaccine.
  Schoolchildren under nine years of age received also one intra-muscular dose of 0.5 ml of varicella vaccine one month after the Meningococcal C vaccine.
  Interventions: Biological: Control vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Influenza vaccine: schoolchidren in the experimental group received IM administered:
  * From 6 to 9 years of age - 2 doses (0.5ml each) of the tri-valent innactivated influenza vaccine - Southern Hemisphere formulation, 2009 - one month apart.
  * 9 years of age and older: one dose (0.5ml) of the tri-valent innactivated influenza vaccine - Southern Hemisphere formulation, 2009 - one month apart.
  Arms: Influenza vaccine
Biological: Control vaccine — Schoolchildren from 6 to 8 years of age:
  - One dose (0.5ml), IM administered, of Meningococcal C conjugate vaccine, and one dose (0.5ml), one month later, of varicella vaccine, IM administered.
  Other Names: Meningococcal C conjugate vaccine; Varicella vaccine
  Arms: Control vaccine

SUMMARY:
Vaccinating schoolchildren against influenza would prevent the disease among non-vaccinated household members.

DETAILED DESCRIPTION:
Children and adolescents play an important role in sustaining the transmission of influenza. Moreover, with the occurrence of influenza in children, there are important socioeconomic consequences to families affected by the disease, related to absenteeism, expenditure on health services and medication use. This study presents an evaluation of direct and indirect effectiveness of influenza vaccination in school age children and their unvaccinated household contacts. It was conducted in 2009, in Sao Paulo - Brazil, through a randomized double-blind community trial, with six months of follow up. For the evaluation of vaccine effectiveness, the influenza vaccine was used for the experimental group, and meningitis conjugate and varicella vaccines for the control group. After vaccination, the volunteers and their families were followed for six months, in order to identify cases of acute respiratory infection (ARI) and to collect biological samples for testing with RT-PCR for diagnosis of influenza.

ELIGIBILITY:
Inclusion Criteria:

* older than six years of age;
* live in the study area;
* parent consent to participate, by signing the Informed Consent Form;
* no history of anaphilaxis or hipersensitivity to eggs or eggs proteins;
* no history no history anaphilaxis or hipersensitivity to any substances;
* no acute disease at the moment of vaccination
* no use of immunesupressant drugs;
* not have received any other vaccine in the previous six months;
* no participation in other clinical trial in the previous six months.

Exclusion Criteria:

* Any condition above mentioned.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1742 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Laboratory confirmed influenza | June 01, 2009 to November 30, 2009
  RT-PCR confirmed influenza in respiratory secretions samples

SECONDARY OUTCOMES:
Acute Repiratory Infection (ARI) | 6 months
  Presence of at least of two symptoms of ARI: fever, cough, sore throat, headache, appetite loss, running nose

OTHER OUTCOMES:
Number of participantes with any adverse event as a measure of safety and tolerability | 30 days after vaccination
  Any solicited or unsolicited adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Expedito J Luna, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Butantan Institute, São Paulo, Brazil